CLINICAL TRIAL: NCT00872807
Title: The Activity School in Finnmark for Overweight and Obese Children and Their Families
Brief Title: The Activity School in Finnmark for Overweight Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: Finnmark Hospital Trust (Other); The Royal Norwegian Ministry of Health (Other); Norwegian Foundation for Health and Rehabilitation (Other); Norwegian Directorate of Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2007/5.2006.3473 (REK); 15873 (NSD) (Other: Norwegian social science data services)
Record Dates: First submitted 2009-03-30; First posted 2009-03-31 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2012-12

CONDITIONS: Obesity; Overweight
Keywords: childhood; therapy; life style; motor activity; obesity; overweight; body mass index; treatment
MeSH Terms: conditions — Obesity; Overweight; Motor Activity | interventions — Population Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group intervention (Experimental): Lifestyle counseling (physical activity and dietary modification) in groups both at the hospital and in their own municipality. They meet a multidisciplinary team, receive organized physical activity in the municipality and are invited to a 3 days camp after 4-6 months.
  Interventions: Behavioral: Lifestyle counseling in groups; Behavioral: Individual intervention
- Individual intervention (Active Comparator): Lifestyle counseling for each separate family practiced by single health professionals both in hospital and municipality. A more conventional model.
  Interventions: Behavioral: Individual intervention

INTERVENTIONS:
Behavioral: Lifestyle counseling in groups — The activity school in Finnmark. Lifestyle counseling (physical activity and dietary modification) in groups both at the hospital and in their own municipality.
  They meet a multidisciplinary team, receive organized physical activity in the municipality and are invited to a 3 days camp after 4-6 months.
  Arms: Group intervention
Behavioral: Individual intervention — Conventional lifestyle counseling individually by single health professionals, both in hospital and in municipality.

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a life style counseling programme designed for overweight and obese children and their parents in groups compared to traditional individual counseling in the pediatric outpatient clinic and the community. The two interventions are both hospital and community based.

DETAILED DESCRIPTION:
Randomized study design with two parallel groups.Active intervention in two years, last follow-up after 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obese.
* BMI > IOTF (International Obesity TaskForce) cut-points 27,5. kg/ m2.

Exclusion Criteria:

* Diseases not compatible with normal physical activity.
* Disorders not compatible with group treatment.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 97 (Actual)
Dates: Start 2009-04; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in Body Mass Index compared to baseline | 3 years
  BMI will be measured at baseline and at 3 months- , 1 year-, 2 year- and 3-year follow-up. Primary measures at 2 years of continuous lifestyle modification. Last measurement at 1 year after last counselling and active treatment has stopped, 3 years from baseline.

SECONDARY OUTCOMES:
Change in Systolic Blood Pressure compared to baseline | 3 years
  Measured with an automated blood pressure monitor at baseline, at 3 months- , 1 year-, 2 year- and 3-year follow-up. Primary measures at the end (2 years) of continuous lifestyle modification. Last measurement at 1 year after last counseling and active treatment has stopped, 3 years from baseline.
Change in Body fat compared to baseline | 3 years
  Measured with bioelectrical impedance analysis at baseline and at 3 months- , 1 year-, 2 year- and 3-year follow-up.Primary measures at 2 years of continuous lifestyle modification. Last measurement at 1 year after last counseling and active treatment has stopped, 3 years from baseline.
Change in activity level / Counts per min compared to baseline | 3 years
  Measured with accelerometers at baseline, 1 year-, 2 year- and 3-year follow-up. Primary measures at 2 years of continuous lifestyle modification. Last measurement at 1 year after last counseling and active treatment has stopped, 3 years from baseline.
Change in Waist circumference compared to baseline | 3 years
  Measured with measuring tape mid-point between the lowest rib and the top of the iliac crest at baseline, 3 months- , 1 year-, 2 year- and 3-year follow-up. Primary measures at 2 years of continuous lifestyle modification. Last measurement at 1 year after last counseling and active treatment stopped, 3 years from baseline.
Change in Homa Score / HOMA IR compared to baseline | 3 years
  Homa score calculated from the cross product of fasting plasma insulin and plasma glucose divided with a factor of 22.5. Fasting plasma insulin and glucose will be measured at baseline, at 1 year-, 2 year- and 3-year follow-up. Primary measures at 2 years of continuous lifestyle modification.Last measurement at 1 year after last counseling and active treatment has stopped, 3 years from baseline.
Change in triceps skinfold compared to baseline | 3 years
  Measured with Holtain Tanner /Whitehouse Skinfold Caliper at baseline,3 months- , 1 year-, 2 year- and 3-year follow-up. Primary measures at 2 years of continuous lifestyle modification.Last measurement at 1 year after last counseling and active treatment has stopped, 3 years from baseline.
Change in self-concept compared to baseline | 3 years
  Measured with SPPC, Self Perception Profile for Children at baseline, at 6 months- , 1 year-, 2 year- and 3-year follow-up. Primary outcome measured at 2 years of continuous lifestyle modification. Last measurement at 1 year after last counseling and active treatment has stopped.
Change in psychiatric health compared to baseline | 3 years
  Measured with Strengths and difficulties Questionnaire ( SDQ-S)at baseline, at 6 months- , 1 year-, 2 year- and 3-year follow-up. Primary measurement at 2 years of continuous lifestyle modification. Last measurement at 1 year after last counseling and active treatment has stopped.
Change in fitness from baseline | 3 years
  Measured with Andersen's test (shuttle test) at baseline, 1 year-, 2 year- and 3-year follow-up. Primary measures at 2 years of continuous lifestyle modification. Last measurement at 1 year after last counseling and active treatment has stopped, 3 years from baseline.
Change in quality of life compared to baseline | 3 years
  Measured with KINDL (Kinder Lebensqualitet Fragebogen) at baseline, 6 months-, 1 year-, 2 year- and 3-year follow-up. Primary measures at 2 years of continuous lifestyle modification. Last measurement at 1 year after last counseling and active treatment has stopped, 3 years from baseline.

OTHER OUTCOMES:
Change in lipid levels compared to baseline | 3 years
  Measurements of total cholesterol, Triglycerides, HDL and LDL at baseline, 1 year-, 2 year- and 3-year follow-up. Primary measures at 2 years of continuous lifestyle modification. Last measurement at 1 year after last counseling and active treatment has stopped, 3 years from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Trond Flægstad, Professor, Study Chair — UNorth Norway
Locations (1):
- Childrens departement Finnmark Hospital, Norway, Hammerfest, Hammerfest, Norway

REFERENCES:
- [Result] Kokkvoll A, Grimsgaard S, Odegaard R, Flaegstad T, Njolstad I. Single versus multiple-family intervention in childhood overweight--Finnmark Activity School: a randomised trial. Arch Dis Child. 2014 Mar;99(3):225-31. doi: 10.1136/archdischild-2012-303571. Epub 2013 Dec 11. PMID 24336385
- [Result] Kokkvoll A, Grimsgaard S, Steinsbekk S, Flaegstad T, Njolstad I. Health in overweight children: 2-year follow-up of Finnmark Activity School--a randomised trial. Arch Dis Child. 2015 May;100(5):441-8. doi: 10.1136/archdischild-2014-307107. Epub 2014 Nov 20. PMID 25414250
- [Derived] Kokkvoll AS, Grimsgaard S, Flaegstad T, Andersen LB, Ball GDC, Wilsgaard T, Njolstad I. No additional long-term effect of group vs individual family intervention in the treatment of childhood obesity-A randomised trial. Acta Paediatr. 2020 Jan;109(1):183-192. doi: 10.1111/apa.14916. Epub 2019 Jul 30. PMID 31240752